CLINICAL TRIAL: NCT06860659
Title: Efficacy of 0.28% Sodium Hyaluronate Eye Drops in Patient with Moderate to Severe Dry Eye : a Randomized Double-blind Controlled Trial
Brief Title: Efficacy of 0.28% Sodium Hyaluronate Eye Drops in Patient with Moderate to Severe Dry Eye
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 67046
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease (DED); Tear Break-Up Time; Tear Disorder; Tear Film Insufficiency; Tear Film Hyperosmolarity; Dry Eye; Hyaluronate; Hyaluronic Acid; Corneal Staining; Quality of Life
Keywords: tear osmolarity; artificial tears; oxford grading scale; DEQS-TH
MeSH Terms: conditions — Dry Eye Syndromes; Xerophthalmia | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The nurse will randomly assign eligible patients to receive either 0.28% sodium hyaluronate eye drops (Vismax®) or 0.18% sodium hyaluronate eye drops (Vislube®) using a computerized randomsation. The nurse will be the only individual informed of the assigned medication and will be responsible for administering the eye drops to the participants.
  Additionally, the nurse will prepare a medication for the patient to take home. TearLAB specialists measured and recorded tear osmolarity before instillation in all cases for 10 minutes, and at 30 and 60 minutes post-instillation. Ophthalmologists evaluated TBUT, ocular surface staining (Oxford grading scale), and the Schirmer I test before instillation for 5 minutes and assessed adverse reactions up to 60 minutes after instillation. Subjects continued treatment for 30 days and were reevaluated during the second visit for OSDI scores, TBUT, the Oxford grading scale, and adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vismax (Experimental): 0.28% Sodium Hyaluronate , preservative free eye drops
  Interventions: Drug: 0.28% Sodium Hyaluronate , preservative free eye drops
- Vislube (Active Comparator): 0.18% Sodium Hyaluronate , preservative free eye drops
  Interventions: Drug: 0.18% Sodium Hyaluronate , preservative free eye drops

INTERVENTIONS:
Drug: 0.28% Sodium Hyaluronate , preservative free eye drops — 0.28% Sodium Hyaluronate , preservative free eye drops
  Arms: Vismax
Drug: 0.18% Sodium Hyaluronate , preservative free eye drops — 0.18% Sodium Hyaluronate , preservative free eye drops
  Arms: Vislube

SUMMARY:
This study aimed to evaluate the efficacy and safety of 0.28% preservative-free SH and 0.18% SH eye drops in patients with dry eye disease. Subjects diagnosed with dry eye disease and meeting the inclusion criteria (Ocular Surface Disease Index (OSDI) score ≥ 23, Fluorescein Tear Breakup Time (TBUT) < 7 seconds were randomized into two groups. Group 1 (42 eyes) received 0.28% SH, and Group 2 (42 eyes) received 0.18% SH, both administered by a nurse. Measurements included tear osmolarity (TearLAB) before instillation and at 0,30 and 60 minutes post-instillation, recorded by a TearLAB specialist. Ophthalmologists assessed TBUT, ocular surface staining (Oxford grading scale), and the Schirmer I test before instillation and evaluated adverse reactions up to 60 minutes post-instillation. Subjects continued treatment for 30 days and were reevaluated during a second visit for OSDI scores, TBUT, the Oxford grading scale, and adverse events. Quality of life score were assessed at before and after treatment for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal 18 year-old
* Ocular Surface Disease Index (OSDI) more than or equal 23
* Oxford grading scale more than or equal 2 (both eye)
* Fluorescein tear break-up time less than 7 seconds (both eyes)
* Willing to being a subject in research.

Exclusion Criteria:

* Diagnosed with other eye diseases that require medication which is not used to treat dry eye, such as Glaucoma
* History of Ocular surgery in previous 3 months or Refractive surgery in previous 6 months
* History of ocular trauma, infection, ocular inflammation which is not involved with dry eye in previous 3 months
* Wear contact lenses
* Allergic to Sodium hyaluronate
* Pregnant or lactation period
* Diagnosed with physical diseases that affect the eyes and cannot yet be controlled, such as uncontrolled DM (Diabetes Mellitus), active autoimmune disease, and systemic neuropathy induced neurotrophic keratopathy. - Continuous use of medications for diseases such as Retinoic acid derivatives, Antihistamines, Cholinergic agents, and Antipsychotic agents which can lead to chronic dry eye
* Incompleted data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-26 (Estimated); Study Completion 2025-06-26 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of 0.28% Sodium Hyaluronate on corneal epithelial healing | 30 days
  The Oxford grading scale was used. This scale consists of six levels: 0, I, II, III, IV, and V, with higher values indicating more severe punctate epithelial erosion.
To examine the effect of 0.28% Sodium Hyaluronate on reducing tear osmolarity | 60 minutes
  Tear osmolarity was monitored before and after the intervention in both arms. Abnormal Tear Osmolarity is defined as a value of ≥ 308 mOsmol/L, measured using the TearLab® system.

SECONDARY OUTCOMES:
3. To study the stability of the tear film following the administration of 0.28% Sodium Hyaluronate | 0 minutes, 60 minutes, and 30 days.
  Fluorescein Tear Break-Up Time (FTBUT) was measured in seconds. Abnormal values are defined as a tear break-up time of ≥ 10 seconds.
To assess dry eye symptoms following the administration of 0.28% Sodium Hyaluronate | 0 minutes and 30 days.
  The Ocular Surface Disease Index (OSDI) was used. The final score is calculated on a scale from 0 to 100, with higher scores indicating greater severity of ocular surface dysfunction.
To assess quality of life following the administration of 0.28% Sodium Hyaluronate | 0 minutes and 30 days.
  The Dry Eye-Related Quality of Life Score (DEQS-Th) was used. The final score is calculated on a scale from 0 to 100, with higher scores indicating greater severity of ocular surface dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Pornlada Sunlakaviset, MD., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, 2, Phayathai Road, Ratchathewi District, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Patient data cannot be disclosed to other researchers because prior consent was not obtained from the patients.

REFERENCES:
- [Background] Tansanguan S, Tananuvat N, Wongpakaran N, Wongpakaran T, Ausayakhun S. Thai version of the dry eye-related quality-of-life score questionnaire: preliminary assessment for psychometric properties. BMC Ophthalmol. 2021 Aug 28;21(1):310. doi: 10.1186/s12886-021-02077-0. PMID 34454466
- [Background] Pattanaphesaj J, Thavorncharoensap M, Ramos-Goni JM, Tongsiri S, Ingsrisawang L, Teerawattananon Y. The EQ-5D-5L Valuation study in Thailand. Expert Rev Pharmacoecon Outcomes Res. 2018 Oct;18(5):551-558. doi: 10.1080/14737167.2018.1494574. Epub 2018 Jul 6. PMID 29958008
- [Background] Prabhasawat P, Tesavibul N, Kasetsuwan N. Performance profile of sodium hyaluronate in patients with lipid tear deficiency: randomised, double-blind, controlled, exploratory study. Br J Ophthalmol. 2007 Jan;91(1):47-50. doi: 10.1136/bjo.2006.097691. Epub 2006 Sep 14. PMID 16973668
- [Background] Troiano P, Monaco G. Effect of hypotonic 0.4% hyaluronic acid drops in dry eye patients: a cross-over study. Cornea. 2008 Dec;27(10):1126-30. doi: 10.1097/ICO.0b013e318180e55c. PMID 19034126
- [Background] Park Y, Song JS, Choi CY, Yoon KC, Lee HK, Kim HS. A Randomized Multicenter Study Comparing 0.1%, 0.15%, and 0.3% Sodium Hyaluronate with 0.05% Cyclosporine in the Treatment of Dry Eye. J Ocul Pharmacol Ther. 2017 Mar;33(2):66-72. doi: 10.1089/jop.2016.0086. Epub 2016 Dec 8. PMID 27929721
- [Background] You IC, Li Y, Jin R, Ahn M, Choi W, Yoon KC. Comparison of 0.1%, 0.18%, and 0.3% Hyaluronic Acid Eye Drops in the Treatment of Experimental Dry Eye. J Ocul Pharmacol Ther. 2018 Oct;34(8):557-564. doi: 10.1089/jop.2018.0032. Epub 2018 Jul 23. PMID 30036099
- [Background] Salzillo R, Schiraldi C, Corsuto L, D'Agostino A, Filosa R, De Rosa M, La Gatta A. Optimization of hyaluronan-based eye drop formulations. Carbohydr Polym. 2016 Nov 20;153:275-283. doi: 10.1016/j.carbpol.2016.07.106. Epub 2016 Jul 29. PMID 27561497
- [Background] Ang BCH, Sng JJ, Wang PXH, Htoon HM, Tong LHT. Sodium Hyaluronate in the Treatment of Dry Eye Syndrome: A Systematic Review and Meta-Analysis. Sci Rep. 2017 Aug 21;7(1):9013. doi: 10.1038/s41598-017-08534-5. PMID 28827614
- [Background] Lopez-de la Rosa A, Pinto-Fraga J, Blazquez Arauzo F, Urbano Rodriguez R, Gonzalez-Garcia MJ. Safety and Efficacy of an Artificial Tear Containing 0.3% Hyaluronic Acid in the Management of Moderate-to-Severe Dry Eye Disease. Eye Contact Lens. 2017 Nov;43(6):383-388. doi: 10.1097/ICL.0000000000000284. PMID 27243353
- [Background] Moschos MM, Chatziralli IP, Sergentanis TN. Viscoat versus Visthesia during phacoemulsification cataract surgery: corneal and foveal changes. BMC Ophthalmol. 2011 Apr 29;11:9. doi: 10.1186/1471-2415-11-9. PMID 21529354
- [Background] Balazs EA. Hyaluronan as an ophthalmic viscoelastic device. Curr Pharm Biotechnol. 2008 Aug;9(4):236-8. doi: 10.2174/138920108785161596. PMID 18691081
- [Background] Shimmura S, Ono M, Shinozaki K, Toda I, Takamura E, Mashima Y, Tsubota K. Sodium hyaluronate eyedrops in the treatment of dry eyes. Br J Ophthalmol. 1995 Nov;79(11):1007-11. doi: 10.1136/bjo.79.11.1007. PMID 8534643
- [Background] Craig JP, Nelson JD, Azar DT, Belmonte C, Bron AJ, Chauhan SK, de Paiva CS, Gomes JAP, Hammitt KM, Jones L, Nichols JJ, Nichols KK, Novack GD, Stapleton FJ, Willcox MDP, Wolffsohn JS, Sullivan DA. TFOS DEWS II Report Executive Summary. Ocul Surf. 2017 Oct;15(4):802-812. doi: 10.1016/j.jtos.2017.08.003. Epub 2017 Aug 8. PMID 28797892
- [Background] Buchholz P, Steeds CS, Stern LS, Wiederkehr DP, Doyle JJ, Katz LM, Figueiredo FC. Utility assessment to measure the impact of dry eye disease. Ocul Surf. 2006 Jul;4(3):155-61. doi: 10.1016/s1542-0124(12)70043-5. PMID 16900272
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342
- [Background] Rolando M, Cantera E, Mencucci R, Rubino P, Aragona P. The correct diagnosis and therapeutic management of tear dysfunction: recommendations of the P.I.C.A.S.S.O. board. Int Ophthalmol. 2018 Apr;38(2):875-895. doi: 10.1007/s10792-017-0524-4. Epub 2017 Apr 10. PMID 28397148
- [Background] Aragona P, Di Stefano G, Ferreri F, Spinella R, Stilo A. Sodium hyaluronate eye drops of different osmolarity for the treatment of dry eye in Sjogren's syndrome patients. Br J Ophthalmol. 2002 Aug;86(8):879-84. doi: 10.1136/bjo.86.8.879. PMID 12140209
- [Background] Fraser JR, Laurent TC, Laurent UB. Hyaluronan: its nature, distribution, functions and turnover. J Intern Med. 1997 Jul;242(1):27-33. doi: 10.1046/j.1365-2796.1997.00170.x. PMID 9260563
- [Background] Sahai A, Malik P. Dry eye: prevalence and attributable risk factors in a hospital-based population. Indian J Ophthalmol. 2005 Jun;53(2):87-91. doi: 10.4103/0301-4738.16170. PMID 15976462
- [Background] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260
- [Background] Dalzell MD. Dry eye: prevalence, utilization, and economic implications. Manag Care. 2003 Dec;12(12 Suppl):9-13. PMID 14723108
- [Background] McCarty CA, Bansal AK, Livingston PM, Stanislavsky YL, Taylor HR. The epidemiology of dry eye in Melbourne, Australia. Ophthalmology. 1998 Jun;105(6):1114-9. doi: 10.1016/S0161-6420(98)96016-X. PMID 9627665
- [Background] Lekhanont K, Rojanaporn D, Chuck RS, Vongthongsri A. Prevalence of dry eye in Bangkok, Thailand. Cornea. 2006 Dec;25(10):1162-7. doi: 10.1097/01.ico.0000244875.92879.1a. PMID 17172891
- See also: Related Info — https://intapi.sciendo.com/pdf/10.5372/1905-7415.0606.134